CLINICAL TRIAL: NCT02044952
Title: Prospective Experimental of Tripterygium Glycoside in the Treatment of Crohn's Disease for Induction Remission
Brief Title: Efficacy and Safety Study of Tripterygium Glycoside in the Treatment of Crohn's Disease for Induction Remission
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhu Weiming (Other)
Responsible Party: Sponsor-Investigator, Zhu Weiming, General Surgery Institute, Jinling Hospital, China
Organization: Jinling Hospital, China (Other)
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CDTW-1
Record Dates: First submitted 2014-01-19; First posted 2014-01-24 (Estimated); Last update posted 2014-01-24 (Estimated); Status verified 2014-01

CONDITIONS: Inflammatory Bowel Diseases; Crohn's Disease; Gastrointestinal Diseases; Digestive System Diseases; Intestinal Diseases
Keywords: Crohn's Disease; mesalazine; Tripterygium Glycosides; induction remission
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Gastrointestinal Diseases; Digestive System Diseases; Intestinal Diseases | interventions — Mesalamine; triptolide; lei gong teng

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mesalazine, Tripterygium glycosides (Experimental): Mesalazine 4g/d and Tripterygium glycosides 2mg/kg/d for 12 weeks
  Interventions: Drug: Mesalazine, Tripterygium glycosides

INTERVENTIONS:
Drug: Mesalazine, Tripterygium glycosides — tripterygium glycosides: 2mg/kg/d, oral Mesalazine: 4g/d, oral
  Other Names: Triptolide; Lei gong teng; Thunder god vine

SUMMARY:
The purpose of this study is to assess the effect and safety of Tripterygium Glycosides in the treatment of Crohn's disease for induction remission and compare the therapeutic effect with patients who received mesalazine.

DETAILED DESCRIPTION:
Crohn's disease is characterized by inflammation and ulceration of the small intestine and colon. Patients commonly experience abdominal pain, diarrhea，malnutrition and malaise which result in decreased quality of life and an increased risk of chronic disability and unemployment.

Tripterygium Glycosides(T2) is a chloroform/methanol extract Tripterygium wilfordii Hook F (TWHF), the traditional Chinese medicine, used in rheumatoid arthritis and nephritis. It has both immune-modulatory and anti-inflammatory activities. Our previous animal studies have revealed that the major component of T2, triptolide, could prevent the development of chronic colitis in interleukin-10 deficient mice. The phase I clinical trial in our institute also demonstrated that T2 is efficient for induction of remission in patients with mild to moderate active crohn's disease. The common adverse effects of T2 are leucopenia, liver renal toxicity, oligospermia and amenorrhea.

The purpose of this study is to assess the effect and safety of Tripterygium Glycosides in the treatment of Crohn's disease for induction remission and compare the therapeutic effect with patients who only received mesalazine.

ELIGIBILITY:
Inclusion Criteria:

* Subjects should have a definitive diagnosis of Crohn's disease, based on WHO criteria.
* Males and females ≥ 18 years old, including women who are not pregnant or lactating at the time of enrollment.
* Subjects should have a CDAI score between 150 to 270 at week 0.
* Able to swallow tablets.
* Are capable of providing written informed consent and obtained at the time of enrollment.
* Willing to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

* Bacterial, viral or other microbial infection(including HIV).
* Orally administered corticosteroids within 3 weeks before enrollment, Inhaled or dermatologic preparations for the treatment of other diseases are acceptable.
* Used of infliximab or immunosuppressant within 2 months before enrollment.
* Previous use of prescription doses of NSAIDs without efficacy.
* Treatment with narcotic pain medications(Anti-diarrheal agents such as loperamide and diphenoxylate are permitted).
* History of pancreatitis, except for subjects with a known but removed cause(such as gallstone pancreatitis).
* History of abnormal liver function tests, including AST or ALT >1.5 times upper limit of normal, alkaline phosphatase >2 times upper limit of normal, total bilirubin >2.5 mg/dL at screening (or within the previous 6 months, if known).
* History of malignancy.
* Women who are pregnant or lactating at the time of enrollment, or who intend to be during the study period.
* Participation in other clinical trial within the past 3 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-05 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Therapeutic effect measured by Crohn's Disease Activity Index (CDAI) | 12 weeks

SECONDARY OUTCOMES:
The Side effects of Tripterygium wilfordii (TW) | 12 weeks
The change of Crohn's Disease Activity Index (CDAI ) | 12Weeks
The change of Simple Endoscopic Score for Crohn's Disease(SES-CD) | 12 Weeks
The change of the Inflammatory Bowel Disease Questionnaire (IBDQ) | 12 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: wei ming zhu, PhD,MD, Principal Investigator — General Surgery Institute, Jinling Hospital
Locations (1):
- General Surgery Institute, Jinling Hospital, Nanjing, Jiangsu, China